CLINICAL TRIAL: NCT06663098
Title: Continued PD-L1 Inhibition With Atezolizumab With Rechallenge Chemotherapy in Patients With Sensitive Relapse SCLC Progressing on First-line Platinum-etoposide Chemotherapy and a PD-L1 Inhibitor: CARRY-ON Study-GOIRC-01-2023
Brief Title: Atezolizumab and Rechallenge Chemotherapy in Relapsed Patients With Extensive-stage Small Cell Lung Cancer (ES-SCLC).
Acronym: CARRY-ON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-01-2023; 2024-511945-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-21; First posted 2024-10-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Keywords: Extensive-stage small cell lung cancer; atezolizumab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): re-challenge chemotherapy plus atezolizumab 1200 mg flat dosing
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV on day 1 of every 21 days, during induction phase and maintenance phase
  Other Names: humanized IgG1 monoclonal antibody against PD-L1
Drug: Carboplatin — AUC 4 or 5, depending on patient's characteristics, on day 1 every 21 days during induction phase
  Other Names: re-challenge chemotherapy
Drug: Etoposide — 80 mg/sqm or 100 mg/sqm, depending on patient's characteristics, on days 1-2-3 of every 21 days
  Other Names: re-challenge chemotherapy

SUMMARY:
The goal of this clinical trial is to learn if a combination of atezolizumab and standard chemotherapy works to treat sensitive Extensive-stage Small Cell Lung Cancer, progressing after first-line of treatment.

The main questions it aims to answer are:

* Does combination of atezolizumab and standard chemotherapy increase overall survival?
* What medical problems do participants have when taking combination of atezolizumab and standard chemotherapy?

Participants will:

* take atezolizumab and standard chemotherapy every 3 weeks for 4 cycles and than atezolizumab every 3 weeks up to 18 cycles.
* visit the clinic once every 3 weeks for checkups and tests
* perform Radiological assessments after 6 weeks and then every 12 weeks to determine response to treatment.

DETAILED DESCRIPTION:
The CARRY-ON study is a multicenter, prospective, open-label single-arm phase II trial, designed to seek for a signal of efficacy of continuing PD-L1 inhibition in patients with sensitive relapse ES-SCLC by adding atezolizumab to rechallenge carboplatin-etoposide chemotherapy. The trial is planned to enroll 142 patients with sensitive relapse ES-SCLC from 25 Italian centers. Sensitive relapse is defined as SCLC relapsed or progressed to first-line chemo-immunotherapy with PD-L1 inhibition (with either atezolizumab or durvalumab) at least 60 days after the last chemotherapy administration. Eligible patients will receive re-challenge chemotherapy (either carboplatin AUC 4 on day 1 plus etoposide 80 mg/m2 days 1-3 or carboplatin AUC 5 on day 1 plus etoposide 100 mg/m2 days 1-3, at investigator's choice) plus atezolizumab 1200 mg flat dosing on day 1 every 3 weeks until PD, unacceptable toxicity or to a maximum of 4 cycles (induction phase) followed by atezolizumab 1200 mg flat dosing every 3 weeks (maintenance phase) until completion of 1 year of maintenance (up to 18 cycles), progressive disease, unacceptable toxicity, patient refusal or loss of clinical benefit (investigator's choice), whichever occur first.

Subjects will attend clinical visits at regular intervals to receive trial treatment and for efficacy and safety assessments. All subjects will be monitored continuously for any AE while on study treatment.

Radiological assessment will be performed by computed tomography (CT) scan at week 6 (± 7 days), at week 12 (± 7 days) and every 12 weeks (± 7 days) thereafter.

The duration of the study is expected to be a maximum of 45 months. The study recruitment period is expected to be approximately 24 months, maximum treatment duration will be 15 months (3 months of induction and 12 months of maintenance), and subsequent survival follow-up will be a maximum of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of small-cell lung cancer (SCLC) (according to WHO classification 2015) confirmed at pathology (histology or cytology).
2. Male or female and ≥ 18 years of age.
3. Life expectancy ≥ 12 weeks.
4. Disease progression at least 60 days after the completion of first-line chemotherapy consisting of at least 4 cycles of platinum-etoposide plus either atezolizumab or durvalumab and have not received any other treatment (except for immunotherapy as maintenance treatment); the 60 day-interval is calculated from the date of the last chemotherapy administration to the date of the first radiologically documented progressive disease.
5. No previous radiotherapy on the only one site disease progression, unless that site had subsequent evidence of progressive disease.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤2.
7. Patients with treated brain metastases (or untreated but asymptomatic) and off steroids or on a stable dose of steroids (≤10 mg of prednisone-equivalent) are also eligible. Radiotherapy must have been completed a minimum of 14 days prior to registration, and patients must have recovered from AEs related to radiotherapy to < grade 1 (except alopecia)
8. For Females: must be postmenopausal (defined as occurring 12 months after last menstrual period) before the screening visit, or are surgically sterile. If they are of childbearing potential, a negative serum pregnancy test prior to study entry has to be documented; furthermore, they agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form (ICF) through 5 months after the last dose of study drug,or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.
9. For Males: even if surgically sterilized (i.e., post-vasectomy status) agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.
10. Normal baseline laboratory values as specified below:

    * Absolute neutrophil count (ANC) ≥1500/mm3
    * Platelet count ≥ 100 x 109/L (≥100,000/μL) without transfusion
    * Hemoglobin ≥ 90 g/L (≥ 9 g/dL); patients may be transfused to meet this criterion.
    * Total bilirubin < 1.5x the institutional upper limit of normal (ULN)
    * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5x the institutional ULN (< 5x if liver function test elevations are due to liver metastases)
    * Creatinine < 1.5x institutional ULN or estimated creatinine clearance using the Cockcroft-Gault formula ≥ 30 mL/minute for patients with creatinine levels above institutional limits
    * For patients not receiving therapeutic anticoagulation: INR and aPTT ≤ 1.5 x ULN
    * Negative HIV test at screening {with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load}
    * Negative hepatitis B surface antigen (HBsAg) test at screening
    * Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

      * Negative total hepatitis B core antibody (HBcAb)
      * Positive total HBcAb test followed by a negative (per local laboratory definition) hepatitis B virus (HBV) DNA testNegative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening The HCV RNA test must be performed for patients who have a positive HCV antibody test.
11. Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before registration, and otherwise noted in other inclusion/exclusion criteria.
12. Recovered (i.e., ≤ grade 1 toxicity) from effects of prior anticancer therapy, except alopecia.
13. Prior radiotherapy is allowed provided that it has been completed more than 2 weeks before starting protocol treatment and patients have recovered from AEs related to radiotherapy to < grade 1
14. Ability to comply with protocol requirements.
15. The patient or the patient's legal representative has to be able to provide written informed consent. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. More than 1 line of prior treatment for ES-SCLC.
2. First-line treatment without either atezolizumab or durvalumab.
3. First-line chemotherapy other than platinum-etoposide.
4. Less than 4 cycles of first-line platinum-etoposide.
5. Presence of resistant relapse (progressive disease within 60 days from the end of first-line chemotherapy) or refractory disease (progressive disease during the first 4 cycles of first-line chemoimmunotherapy).
6. Symptomatic brain metastases or spinal cord compression (CT or MRI of the head is required within 4 weeks prior to randomization)requiring immediate radiotherapy for palliation. Patients with treated brain metastases (or untreated but asymptomatic) and off steroids or on a stable dose of steroids (≤10 mg of prednisone-equivalent) are also eligible provided that all of the following criteria are met:

   * If treated, at least 14 days between the end of stereotactic radiotherapy or whole brain radiotherapy and initiation of study treatment and recovery from AEs related to radiotherapy to ≤ grade 1 (except alopecia), or at least 28 days between neurosurgical resection and initiation of study treatment;
   * Anticonvulsant therapy at a stable dose is permitted;
   * Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla or spinal cord);
   * There is no evidence of interim intracranial progression between completion of CNS directed therapy (if administered) and initiation of study treatment.
7. Evidence of leptomeningeal disease.
8. Any comorbid condition or unresolved toxicity that would preclude administration of second-line chemotherapy.
9. Patient has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines and COVID vaccines that do not contain live virus are permitted. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
10. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment except for PD-L1 inhibitor maintenance as part of first-line treatment.
11. Any condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of registration . The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection);
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent;
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
12. Diagnosed with or treated for another malignancy within 3 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type may be enrolled in the study if they have undergone complete resection and no evidence of active disease is present.
13. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment other than those in the present study. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
14. Treatment with any other investigational agent within 30 days prior to starting study treatment, or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
15. Infection requiring intravenous antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
16. Prior allogeneic stem cell or solid organ transplantation.
17. For female subjects: positive serum pregnancy test, pregnancy, or breastfeeding.
18. Surgery within 4 weeks (or 2 weeks for a minor surgery) before study enrolment and not fully recovered to baseline or to a stable clinical status. Insertion of a vascular device is allowed.
19. Patients who experienced medically significant or NCI CTCAE Grade 3 or higher toxicities in response to first-line immunotherapy
20. Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | through study completion, an average of 1 year
  overall survival (OS), defined as the time from the date of registration to the date of death from any cause. Patients still alive at the time of analysis are censored at the last time they are known to be alive.

SECONDARY OUTCOMES:
frequency of adverse events | 30 days post last dose of study drug
  Toxicity will be assessed in the mITT population. Descriptive tables will be produced which provide the worst degree of toxicity measured over all cycles according to the NCI-CTCAE version 5.0
Progression Free Survival | through study completion, an average of 6 months
  Progression Free Survival (PFS) defined as the time from the patient registration to the evidence of progressive disease, or death, or the last date the patient was known to be progression-free and alive.
Objective response rate | through study completion, an average of 1 year
  Objective response rate (ORR) is calculated as the sum of RECIST v1.1-defined CR and PR out of the number of assessable patients with measurable disease at baseline.

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - Centro di Riferimento Oncologico di Aviano (CRO) IRCCS, Aviano (PN)
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - IRCCS Azienda Ospedaliero_Universitaria di Bologna, Bologna
  - UOC Medicina Oncologica, Carpi
  - ASST Cremona, Cremona
  - Azienda Ospedaliera S. Croce e Carle di Cuneo, Cuneo
  - AOU Careggi, Florence
  - Azienda USL Toscana nord-ovest Ospedale Versilia, Lido di Camaiore
  - Azienda USL Toscana Nord Ovest - Ospedale San Luca, Lucca
  - Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori (IRST) "Dino Amadori", Meldola (FC)
  - IRCCS Ospedale San Raffaele, Milan
  - AOU Policlinico di Modena, Modena
  - ASST San Gerardo dei Tintori Foundation, Monza
  - AORN A. Cardarelli, Napoli
  - AOU San Luigi Gonzaga, Orbassano (TO)
  - Istituto Oncologico Veneto, Padua
  - UOC di Oncologia Medica, Parma
  - Azienda Ospedaliera Santa Maria della Misericordia, Perugia
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Fondazione Policlinico Universitario A.Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - AOU Sassari, Sassari
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Azienda Sanitaria Universitaria Friuli Centrale - P.O. Santa Maria della Misericordia, Udine
  - AOU Integrata di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansfield AS, Kazarnowicz A, Karaseva N, Sanchez A, De Boer R, Andric Z, Reck M, Atagi S, Lee JS, Garassino M, Liu SV, Horn L, Wen X, Quach C, Yu W, Kabbinavar F, Lam S, Morris S, Califano R. Safety and patient-reported outcomes of atezolizumab, carboplatin, and etoposide in extensive-stage small-cell lung cancer (IMpower133): a randomized phase I/III trial. Ann Oncol. 2020 Feb;31(2):310-317. doi: 10.1016/j.annonc.2019.10.021. Epub 2019 Dec 9. PMID 31959349
- [Background] Zitvogel L, Galluzzi L, Smyth MJ, Kroemer G. Mechanism of action of conventional and targeted anticancer therapies: reinstating immunosurveillance. Immunity. 2013 Jul 25;39(1):74-88. doi: 10.1016/j.immuni.2013.06.014. PMID 23890065
- [Background] Li L, Liu T, Liu Q, Mu S, Tao H, Yang X, Li Y, Xiong Q, Wang L, Hu Y. Rechallenge of immunotherapy beyond progression in patients with extensive-stage small-cell lung cancer. Front Pharmacol. 2022 Sep 6;13:967559. doi: 10.3389/fphar.2022.967559. eCollection 2022. PMID 36147357
- [Background] Spagnolo F, Boutros A, Cecchi F, Croce E, Tanda ET, Queirolo P. Treatment beyond progression with anti-PD-1/PD-L1 based regimens in advanced solid tumors: a systematic review. BMC Cancer. 2021 Apr 17;21(1):425. doi: 10.1186/s12885-021-08165-0. PMID 33865350
- [Background] Ardizzoni A, Tiseo M, Boni L. Validation of standard definition of sensitive versus refractory relapsed small cell lung cancer: a pooled analysis of topotecan second-line trials. Eur J Cancer. 2014 Sep;50(13):2211-8. doi: 10.1016/j.ejca.2014.06.002. Epub 2014 Jun 26. PMID 24981975
- [Background] Baize N, Monnet I, Greillier L, Geier M, Lena H, Janicot H, Vergnenegre A, Crequit J, Lamy R, Auliac JB, Letreut J, Le Caer H, Gervais R, Dansin E, Madroszyk A, Renault PA, Le Garff G, Falchero L, Berard H, Schott R, Saulnier P, Chouaid C; Groupe Francais de Pneumo-Cancerologie 01-13 investigators. Carboplatin plus etoposide versus topotecan as second-line treatment for patients with sensitive relapsed small-cell lung cancer: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2020 Sep;21(9):1224-1233. doi: 10.1016/S1470-2045(20)30461-7. PMID 32888454
- [Background] Frampton JE. Atezolizumab: A Review in Extensive-Stage SCLC. Drugs. 2020 Oct;80(15):1587-1594. doi: 10.1007/s40265-020-01398-6. PMID 32990939
- [Background] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- [Background] Liu SV, Reck M, Mansfield AS, Mok T, Scherpereel A, Reinmuth N, Garassino MC, De Castro Carpeno J, Califano R, Nishio M, Orlandi F, Alatorre-Alexander J, Leal T, Cheng Y, Lee JS, Lam S, McCleland M, Deng Y, Phan S, Horn L. Updated Overall Survival and PD-L1 Subgroup Analysis of Patients With Extensive-Stage Small-Cell Lung Cancer Treated With Atezolizumab, Carboplatin, and Etoposide (IMpower133). J Clin Oncol. 2021 Feb 20;39(6):619-630. doi: 10.1200/JCO.20.01055. Epub 2021 Jan 13. PMID 33439693
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Dingemans AC, Fruh M, Ardizzoni A, Besse B, Faivre-Finn C, Hendriks LE, Lantuejoul S, Peters S, Reguart N, Rudin CM, De Ruysscher D, Van Schil PE, Vansteenkiste J, Reck M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Small-cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up☆. Ann Oncol. 2021 Jul;32(7):839-853. doi: 10.1016/j.annonc.2021.03.207. Epub 2021 Apr 20. No abstract available. PMID 33864941
- [Background] Yang S, Zhang Z, Wang Q. Emerging therapies for small cell lung cancer. J Hematol Oncol. 2019 May 2;12(1):47. doi: 10.1186/s13045-019-0736-3. PMID 31046803